CLINICAL TRIAL: NCT00483977
Title: A 2 Week, Randomized, Double Blind, Placebo And Positive Controlled, Parallel Group, Multicentre Study To Assess The Efficacy And Tolerability Of PF-00592379 In Patients With Moderate To Severe Pain Due To Osteoarthritis
Brief Title: A 2 Week Blinded Study For Pain Due To Arthritis Of The Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Met criteria for study futility at interim analysis
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7771010
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxycodone (Active Comparator)
  Interventions: Drug: Oxycodone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-00592379 (Experimental)
  Interventions: Drug: PF-000592379

INTERVENTIONS:
Drug: Oxycodone — Oxycodone: oral controlled release, 20 mg, twice a day for 2 weeks
  Arms: Oxycodone
Drug: Placebo — Placebo: oral for 2 weeks.
  Arms: Placebo
Drug: PF-000592379 — PF-00592379: oral, 30 mg, once a day for 2 weeks
  Arms: PF-00592379

SUMMARY:
The primary aim is to assess if PF-00592379 is able to reduce pain in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race
* Between the ages of 18 and 75 years
* Knee Pain due to osteoarthritis

Exclusion Criteria:

* Pregnant
* Participation in a clinical trial for an investigational drug and/or agent within 30 days prior to baseline
* History of malignancy, convulsions, chronic infections, arthroscopy of the worst knee within the past year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the pain score averaged over the last week of treatment | 2 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) pain score - change from baseline to end of treatment | 2 weeks
Patient Global Impression of Change | 2 weeks
Patients Global Assessment of Osteoarthritis | 2 weeks
Pharmacokinetic trough levels | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Fair Oaks, California
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Richmond, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7771010&StudyName=A%202%20Week%20Blinded%20Study%20For%20Pain%20Due%20To%20Arthritis%20Of%20The%20Knee.